CLINICAL TRIAL: NCT00587548
Title: Intraoperative Gamma Probe Localization of the Ureter
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided not pursue the study
Sponsor: Mayo Clinic (Other)
Responsible Party: Manpreet Grewal, M.D., Mayo Clinic Jacksonville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 79-06; MCJ092006
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Abdominal Surgery
Keywords: locate the ureters during abdominal surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Localizing the ureters during surgery — One-time injection 4.5mCi of 99mTechnetium labeled diethylene-triamine-penta acetate (DTPA) prior to the time of ureteral localization. The Neoprobe 2000 gamma probe will be utilized for ureter location.
  Other Names: 4.5cmCi 99mTechnetium labeled diethylene-triamine-penta acetate (DTPA); Neoprobe 2000 gamma probe

SUMMARY:
This study is being done to find a different way to identify the ureters during an abdominal operation.

During some operations, the operating physician must identify where the ureters are to prevent injury to them. Typically, the surgeon calls the urologist to thread a small scope with a camera into the urethra (where the urine comes out) to place a wire into each of the two ureters to locate them. Instead of this procedure, we will inject a small amount of a radioactive chemical dye (TC99-DTPA)through a vein in your arm. The ureters can then be detected by a hand held probe called the 'gamma probe.' The TC99-DTPA dye passes through the body and is excreted through the urine. The goal of this study is that this probe will alert the physician when it placed directly over the ureters since the TC99-DTPA dye will highlight the ureters as the flow of urine goes through them.

DETAILED DESCRIPTION:
The patient population includes those that are undergoing an elective, open, abdominal surgery.

The patient will receive, on average, 4.5mCi of Technetium labeled diethylene-triamine-penta acetate (DTPA) prior to the time of ureteral localization. The Neoprobe 2000 gamma probe will be placed on the field in sterile fashion in a manner similar to that which is performed during a minimally invasive parathyroidectomy or sentinel lymph node biopsy. The surgery will continue until the surgical team feels the time is appropriate for each ureter to be identified. At this point, the surgical team will use the gamma probe to localize the ureter and the attending physician will note either, "yes" or, "no" to their feeling is that they have correctly identified or did not identify each ureter. The surgical team will know that the ureter has been correctly identified when gentle manipulation of the tissue with forceps produces a "vermicular contraction" of the tubular structure suspected to be the ureter. No other tissue and/or structure produces this classic type of contraction. Background gamma counts, gamma counts over the ureter, and time between Tc-DTPA injection and ureteral localization will be recorded for each ureter sought. If the ureter cannot be localized with this technique, and the surgical team feels that it is imperative that the ureters be identified, then the attending surgeon may request a urologist to place stents in the standard, usual fashion.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to informed consent.
* Patients undergoing elective, open, abdominal surgery
* 18 years or older
* Normal renal function defined by a serum creatinine less than 1.5mg/dL

Exclusion Criteria:

* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
If gamma probe localization of the ureters is possible, the need for ureteral stent placement could be obviated. | Intraoperative procedure

CONTACTS AND LOCATIONS:
Overall Officials: Manpreet Grewal, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Jacksonville, Jacksonville, Florida, United States